CLINICAL TRIAL: NCT07195110
Title: Prevalence of Periodontal Disease Among Egyptian Patients With Multiple Sclerosis S: A Cross Sectional Study
Brief Title: Prevalence of Periodontitis in Egyptian Multiple Sclerosis Patients.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Mohamed wageh Eltonsy, Principal investigator, Cairo University
Other Study IDs: PER4-1-2
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis (MS); Periodontal Diseases
MeSH Terms: conditions — Multiple Sclerosis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the association between multiple sclerosis and periodontal disease in a sample of Egyptian population

The main question it aims to answer is:

• Is there an association between MS and periodontal disease Participants already diagnosed with multiple sclerosis. A conventional oral examination will be held on a dental unit, filling charts and patients' acceptance to participate in the survey.

DETAILED DESCRIPTION:
Periodontal disease is a chronic inflammatory condition leading to progressive destruction of the supporting structures of the teeth. Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system that may share common inflammatory pathways with periodontal disease. Recent evidence suggests that systemic inflammation may influence the severity and progression of both conditions.

This study will recruit participants already diagnosed with MS and assess their periodontal status using standard clinical parameters, including clinical attachment loss (CAL), probing pocket depth, and bleeding on probing measured at six sites per tooth using a periodontal probe. Data will be collected through a conventional oral examination in a dental unit, and results will be compared to evaluate the prevalence and potential association between MS and periodontal disease within this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MS
* Adult patients ≥ 18 years old.
* Patients providing an informed consent

Exclusion Criteria:

* Periodontal therapy within the last 3 months.
* Having surgical therapy or undergoing orthodontic treatment
* Smokers
* Pregnant females
* Patients with systemic condition know to impact the periodontal condition other than MS (eg. Diabetes Mellitus)
* Patients having more than 5 lost teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients to be recruited and selected from sheikh Zayed Al-Nahayan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 293 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periodontal disease as assessed by clinical periodontal parameters ( clinical attachment loss )within the study population. | Baseline
  CAL will be measured as the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket using a periodontal probe at six sites per tooth. Mean CAL will be calculated for each participant to assess periodontal tissue destruction.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and limitations in data-sharing infrastructure. Only aggregate study results will be published and made publicly available.